CLINICAL TRIAL: NCT01742689
Title: Assessment of Analgesic Efficacy of Intranasal Desmopressin in the Treatment of Acute Pain in Patients With Renal Colic
Brief Title: Analgesic Efficacy of Intranasal Desmopressin in Acute Renal Colic
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91/130/569
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Renal Colic; Pain
Keywords: Renal colic; Pain; Desmopressin; Urinary obstruction; Indomethacin
MeSH Terms: conditions — Renal Colic; Pain | interventions — Deamino Arginine Vasopressin; Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desmopressin intranasal spray (Experimental): Patients in this arm will receive 40 microgram desmopressin intranasal spray & 100 milligram indomethacin suppository
  Interventions: Drug: Desmopressin intranasal spray; Drug: Indomethacin suppository
- Placebo intranasal spray (Placebo Comparator): Patients in this group will receive placebo nasal spray & 100 milligram indomethacin suppository
  Interventions: Drug: Placebo intranasal spray; Drug: Indomethacin suppository

INTERVENTIONS:
Drug: Desmopressin intranasal spray — 10 microgram per puff, 40 microgram is Descript
  Other Names: DDAVP, DesmoMelt, Stimate, Minirin,Desmex
  Arms: Desmopressin intranasal spray
Drug: Placebo intranasal spray — Saline spray identical to desmopressin, administered as 4 sprays
  Arms: Placebo intranasal spray
Drug: Indomethacin suppository — Indomethacin suppository 100 milligram single dose
  Other Names: Indocin; Indocid; Indochron; INDOMET

SUMMARY:
In this study we will compare pain intensity and side effects at different time points after the intranasal administration of desmopressin or placebo in patients with acute renal colic pain.

DETAILED DESCRIPTION:
Obstruction of the urinary tract can increase pelvi-ureteric pressure and thus cause renal colic pain, which can be very severe. Conventional therapy consists of non-steroidal anti-inflammatory drugs (NSAIDs) and opioids. NSAIDs have many side effects and opioids are not always available. In addition, the intravenous form of NSAIDs is not routinely available in Iran, and the drug is mainly used in the form of suppository. Due to these reasons, research on newer replacement therapies with fewer side effects is necessary. Desmopressin intranasal spray has already been shown to be partially effective in renal colic pain in a few studies. Due to its lower side effects, we decided to conduct a clinical trial with desmopressin to evaluate pain relief in renal colic. In this study, eighty-eight patients with acute renal colic pain, referring to Imam Khomeini Hospital in Tehran, will be randomly allocated to receive either intranasal desmopressin or placebo. Both groups will also receive 100 milligram indomethacin suppository. Pain intensity will be assessed and recorded using a verbal numeric rating scale, before nasal spray, and in minutes 5, 10, 15, 30, 45 and 60 after receiving the allocated treatment. Possible side effects will also be asked and recorded. The patient and the investigator responsible for recording pain intensity will not be aware of the administered drug. The results will be compared before and after treatment in each group, using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Age: 15 to 65 years
* Pain intensity of at least 3
* Clinical diagnosis of renal colic

Exclusion Criteria:

* History of hypertension
* History of acute myocardial ischemia
* History of hyponatremia
* Presence of acute rhinitis and flu
* Coagulopathy or anticoagulant therapy
* History of peptic ulcer disease, asthma, renal failure, severe liver failure
* Analgesic use over 4 hours ago
* Taking seizure medications (such as carbamazepine)
* Taking any of the following drugs: chlorpropamide, warfarin, clofibrate , epinephrine, Fludrocortisone, heparin, lithium, alcohol

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | baseline till one hour
  Changes in pain intensity using a verbal numeric rating scale

SECONDARY OUTCOMES:
Side effects | One hour
  Any perceived side effects reported by the patient, including dry mouth, nausea, and drowsiness.

OTHER OUTCOMES:
Use of opioid as a rescue drug | One hour
  Whether or not the patient care team had to administer opioids due to uncontrolled pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jalili, MD, Study Chair — Tehran University of Medical Sciences; Mohammadreza Hedayatshodeh, MD, Study Director — Tehran University of Medical Sciences
Locations (2):
- Iran (2):
  - Imam Khomeini General Hospital, Tehran, Tehran Province
  - Shariati Hospital, Tehran, Tehran Province

REFERENCES:
- [Background] Roshani A, Falahatkar S, Khosropanah I, Roshan ZA, Zarkami T, Palizkar M, Emadi SA, Akbarpour M, Khaki N. Assessment of clinical efficacy of intranasal desmopressin spray and diclofenac sodium suppository in treatment of renal colic versus diclofenac sodium alone. Urology. 2010 Mar;75(3):540-2. doi: 10.1016/j.urology.2008.05.053. Epub 2009 Dec 4. PMID 19962730
- [Background] Lopes T, Dias JS, Marcelino J, Varela J, Ribeiro S, Dias J. An assessment of the clinical efficacy of intranasal desmopressin spray in the treatment of renal colic. BJU Int. 2001 Mar;87(4):322-5. doi: 10.1046/j.1464-410x.2001.00068.x. PMID 11251523